CLINICAL TRIAL: NCT01524705
Title: FLAT-SUGAR: FLuctuATion Reduction With inSULin and Glp-1 Added togetheR
Brief Title: FLuctuATion Reduction With inSULin and Glp-1 Added togetheR (FLAT-SUGAR)
Acronym: FLAT-SUGAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eli Lilly and Company (Industry); Sanofi (Industry); Astra Zeneca, Bristol-Myers Squibb (Other); DexCom, Inc. (Industry); Bayer (Industry); Becton, Dickinson and Company (Industry); Medicomp (Unknown); University of Texas (Other); US Department of Veterans Affairs (U.S. Federal Agency); Biomedical Research Institute of New Mexico (Other)
Responsible Party: Principal Investigator, Jeff Probstfield, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42178
Record Dates: First submitted 2012-01-17; First posted 2012-02-02 (Estimated); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes
Keywords: Pilot Study; Prospective Randomized Trial; Comparative Effectiveness; Glycemic Variability; insulin glargine; exenatide; basal insulin; bolus insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Metformin; Insulin Aspart; Insulin Lispro; Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin Glargine, metformin, exenatide (Experimental): Approximately 60 Type 2 diabetes mellitus (DM) participants will be instructed on an American Heart Association/American Diabetes Association (AHA/ADA) meal plan. Insulin Glargine, metformin and exenatide will used as a combination strategy to control individual glycosylated hemoglobin level (HbA1Cs) between 6.7 and 7.3% throughout the trial. The use of exenatide makes this the intervention arm
  Interventions: Drug: Insulin Glargine; Drug: Metformin; Drug: Exenatide
- glargine, metformin, prandial insulin (Active Comparator): Approximately 60 type 2 DM participants will be instructed in AHA/ADA meal plan. Insulin Glargine, metformin and one of 3 prandial insulins will be used as combination strategy to control individual HbA1Cs between 6.7 and 7.3%. Prandial Insulins (aspart, glulisine or lispro). The use of the short acting insulins make this the control arm
  Interventions: Drug: Insulin Glargine; Drug: Metformin; Drug: Prandial insulin

INTERVENTIONS:
Drug: Insulin Glargine — Glargine-injectable, variable, once daily (QD), 6 months
  Other Names: Basal insulin
Drug: Metformin — Metformin-oral, up to 1000mg, twice daily (BID), 6 months
  Other Names: Generic metformin
Drug: Prandial insulin — Aspart or glulisine or lispro
  Other Names: Aspart or glulisine or lispro
  Arms: glargine, metformin, prandial insulin
Drug: Exenatide — Injectable, 5mcg, twice daily (BID), 6 months
  Other Names: Glucagon-like polypeptide-1-agonist (GLP-1-agonist); Byetta
  Arms: Insulin Glargine, metformin, exenatide

SUMMARY:
Results of recent studies using standard long and short acting insulin therapy (Basal - Bolus or BBI) in type 2 diabetes mellitus (T2DM) have not shown benefits to lower risks for heart attacks, strokes, or eye, nerve and kidney problems. Some studies also show a long time between the start of treatment and signs of benefit. This has led to a review of current ways to normalize blood glucose control with basal bolus insulin and how to make blood glucose better. Improving blood sugar with insulin therapy usually causes weight gain, more high sugar levels after meals, and more low blood sugars. Early studies suggest that when people take long-acting insulin and metformin, they have fewer blood sugar extremes when they also take a new type of medicine called glucagon-like polypeptide-1 (GLP-1) agonist named exenatide (Byetta), instead of meal-time insulin. This means there might be a better way to treat Type 2 diabetes.

Participants are asked to take part in an eight month study to find out if middle-aged and older people with Type 2 diabetes who have added risk factors for heart disease can even out their blood sugar levels. They will start on long-acting insulin, mealtime insulin, and metformin, if they are not already on these medications. Their kidney function tests must be normal and they must not be allergic to metformin. Then, after a 2 month run-in phase, they must be willing to be assigned by chance into one of two groups. This means that they will have a 50/50 chance (like flipping a coin) of being in either group. Half of them will be started on the new medicine known as Byetta rather than the meal-time insulin and the other half will remain on the meal-time insulin during the next 6 months (26 weeks) to see which group has more steady blood sugars. They will be asked to use a continuous blood sugar monitoring system called DexCom. A sensor is inserted under the skin in the same areas the insulin is injected. The DexCom can check their blood sugars 24 hours of the day and night and will be worn until 7 days of recordings are collected. In the same 7 day period, they will also be asked to wear a Holter or Telemetry monitor that will record their heart beats and rhythm which will be compared to the blood sugar readings. They will also use home glucose meters to check their glucose levels about 3 to 4 times a day. The study will take place at 12 centers in the United States and enroll about 120-130 people.

DETAILED DESCRIPTION:
Recent medical endpoint studies employing conventional basal bolus insulin therapy (BBI) in type 2 diabetes mellitus (T2DM) have been disappointing, showing either inconsistent or no effect of treatments on risks for micro- or macro-vascular events, or a long interval between treatment initiation and evidence of clinical benefit. In fact, one trial has suggested that treating glycosylated hemoglobin (HbA1C) to lower targets may even lead to harm. This has raised the possibility that more aggressive glucose lowering approaches lead to harm that overwhelms benefit in those with T2DM. Potential explanations for these results include three closely related physiologic processes: glycemic variability, weight gain and hypoglycemia. Too much variability of glucose, especially post-prandial hyperglycemia, poses the dilemma of how to achieve near-normal mean glucose and HbA1C levels without causing insulin-induced hypoglycemia and/or weight gain. All three of these processes have been linked to worsening systemic inflammation and oxidative stress, and to increased renal and cardiovascular risks.

Fortunately, new tools are available that allow us to assess the severity of glycemic variability (continuous glucose monitoring, or CGM), and to investigate the mechanisms through which it may lead to cardiovascular risk (e.g., systemic inflammation and oxidative stress, sensitive measures of diabetic renal disease, and Holter or Telemetry monitoring for hypoglycemia-induced arrhythmias). In addition, preliminary studies have suggested that replacement of rapid-acting analogue (RAA) in traditional BBI with the glucagon-like polypeptide-1 (GLP-1) agonist, exenatide, may substantially reduce glycemic variability without a strong tendency to increase body weight or hypoglycemia.

This research trial, "FLuctuATion reduction with inSUlin and Glp-1 Added togetheR (FLAT-SUGAR)", by using these new methods to optimize glycemic control while limiting unwanted adverse effects, will be a definitive comparative effectiveness trial. This trial is designed to address the following primary hypothesis:

In middle aged and older individuals with T2DM and additional risk factors for cardiovascular disease, and on a background therapy of basal insulin (insulin glargine) and metformin, the addition of the GLP-1 analogue, exenatide, reduces glycemic variability more than the addition of a rapid-acting-analogue (RAA) (insulin aspart, insulin glulisine or insulin lispro) during an active treatment period of 26 weeks.

The primary outcome measure will be the change in the coefficient of variation of continuous glucose readings, as assessed by CGM. Importantly, FLAT-SUGAR will plan, a priori, to assess glycemic variability using CGM. Secondary trial goals will be to explore potential between-group differences in complications that may result from glycemic variability, including hypoglycemia, systemic inflammation and oxidant stress, diabetic renal disease, weight gain and cardiac arrhythmias. If, as we expect, FLAT-SUGAR demonstrates that CGM provides objective verification of reduced glycemic variability in T2DM with the new GLP-1 agonist-based regimen, the main goal of the trial will be accomplished. If reduced variability is associated with lower risks of adverse events of inflammation, albuminuria progression, weight gain, hypoglycemia, and/or cardiac arrhythmia, a long term clinical comparative effectiveness trial powered to evaluate medical outcomes will be justified.

In order to conduct FLAT-SUGAR, a randomized, controlled, multicenter, open-label investigator-initiated trial, the primary funding is supported by Sanofi-Aventis US with donations of other medications and devices by several other companies. The Sponsor-Investigator is the University of Washington, which will also be the Operation Center (OC).The Data Center (DC) is the University of Texas at Houston School of Public Health. There will be 12 clinical sites with diabetes and CGM expertise to screen and enroll qualified participants for approximately 8-10 weeks of a run-in period, then ultimately randomize, and follow 120 total participants for an active treatment period of 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. T2DM for >12 months defined according to current ADA criteria
2. C-peptide >0.5 ng/mL-after informed consent has been signed, samples will be drawn fasting and sent to a central lab
3. Participants must be on insulin therapy. Diabetes, Blood Pressure & Lipid therapy must be stable (in both dose and agent) for ≥3 months (dose of any 1 drug has not changed by more than 2-fold, & new agents not been added within the previous 3 months)
4. HbA1c 7.5-8.5% for enrollment
5. Age at enrollment (screening): 40-75 years (inclusive) when there is a history of cardiovascular disease (defined in 'a'), or 55 to 75 years (inclusive) when there is not a history of cardiovascular disease but 2 or more risk factors (with or without treatment) are present (defined in 'b')

   a) Established cardiovascular disease defined as presence of one of the following: i. Previous myocardial infarction (MI). (most recent must be > 3 months prior enrollment) ii. Previous stroke. (most recent must be >3 months prior enrollment) iii. History of coronary revascularization (e.g., coronary artery bypass graft surgery, stent placement, percutaneous transluminal coronary angioplasty, or laser atherectomy)(most recent must be > 3 months prior enrollment) iv. History of carotid or peripheral revascularization (e.g., carotid endarterectomy, lower extremity atherosclerotic disease atherectomy, repair of abdominal aortic aneurysm, femoral or popliteal bypass). (most recent must be >3 months prior enrollment) v. Angina with either ischemic changes on a resting ECG, or ECG changes on a graded exercise test (GXT), or positive cardiac imaging study vi. Ankle/brachial index <0.9 vii. LVH with strain by ECG or ECHO viii. >50% stenosis of a coronary, carotid, renal or lower extremity artery. ix. Urine albumin to urine creatinine ratio of >30 mg albumin/g creatinine in 2 samples, separated by at least 7 days, within past 12 months) [Target of 50% of study cohort] or b) Increased CVD risk defined as presence of 2 or more of the following: i. Untreated LDL-C >130 mg/dL or on lipid treatment ii. Low HDL-C (<40 mg/dL for men and <50 mg/dL for women) iii. Untreated systolic BP >140 mm Hg, or on antihypertensive treatment iv. Current cigarette smoking v. Body mass index 25-45 (Asian populations 23-45) kg/m2
6. No expectation that participant will move out of clinical center area during the next 8 months, unless move will be to an area served by another trial center
7. Ability to speak & read English

Exclusion Criteria:

1. The presence of a physical disability, significant medical or psychiatric disorder; substance abuse or use of a medication that in the judgment of the investigator will affect the use of CGM, wearing of the sensors, Holter or Telemetry monitor, complex medication regimen, or completion of any aspect of the protocol
2. Cannot have had any cardiovascular event or interventional procedure, (MI, Stroke or revascularization) or been hospitalized for unstable angina within the last 3 months
3. Inability or unwillingness to discontinue use of acetaminophen products during CGM use
4. Inability or unwillingness to discontinue use of all other diabetes agents other than insulin & metformin during trial (including insulin pump participants who will need to convert to BBI)
5. Intolerance of metformin dose <500 mg/day
6. Inability or unwillingness to perform blood glucose testing a minimum of 3 times/per day
7. Creatinine level ≥1.5 for males or 1.4 for females
8. ALT level ≥ 3 times upper limit of normal
9. Current symptomatic heart failure, history of NYHA Class III or IV congestive heart failure at any time, or ejection fraction (by any method) < 25%
10. Inpatient psychiatric treatment in the past 6 months
11. Currently participating in an intervention trial
12. Chronic inflammatory diseases, such as collagen vascular diseases or inflammatory bowel disease
13. History of pancreatitis
14. BMI >45kg/m2
15. For females, pregnant or intending to become pregnant during the next 7 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Probstfield, MD, Principal Investigator — Professor of Medicine, University of Washington
Locations (12):
- United States (12):
  - So Calif. Permanente Medical Group, San Diego, California
  - University of Miami, Miami, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Joslin Diabetes Center, Boston, Massachusetts
  - International Diabetes Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Kaledia Health of Western New York, Buffalo, New York
  - Diabetes Care Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Vermont, Colchester, Vermont
  - University of Washington, Seattle, Washington
  - Washington State University Spokane, College of Pharmacy Spokane WA 99202 USA, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data available from the authors
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Written request to the investigators

REFERENCES:
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Background] Duckworth W, Abraira C, Moritz T, Reda D, Emanuele N, Reaven PD, Zieve FJ, Marks J, Davis SN, Hayward R, Warren SR, Goldman S, McCarren M, Vitek ME, Henderson WG, Huang GD; VADT Investigators. Glucose control and vascular complications in veterans with type 2 diabetes. N Engl J Med. 2009 Jan 8;360(2):129-39. doi: 10.1056/NEJMoa0808431. Epub 2008 Dec 17. PMID 19092145
- [Background] Davi G, Ciabattoni G, Consoli A, Mezzetti A, Falco A, Santarone S, Pennese E, Vitacolonna E, Bucciarelli T, Costantini F, Capani F, Patrono C. In vivo formation of 8-iso-prostaglandin f2alpha and platelet activation in diabetes mellitus: effects of improved metabolic control and vitamin E supplementation. Circulation. 1999 Jan 19;99(2):224-9. doi: 10.1161/01.cir.99.2.224. PMID 9892587
- [Background] Tannock LR, O'Brien KD, Knopp RH, Retzlaff B, Fish B, Wener MH, Kahn SE, Chait A. Cholesterol feeding increases C-reactive protein and serum amyloid A levels in lean insulin-sensitive subjects. Circulation. 2005 Jun 14;111(23):3058-62. doi: 10.1161/CIRCULATIONAHA.104.506188. Epub 2005 Jun 6. PMID 15939816
- [Background] Festa A, D'Agostino R Jr, Howard G, Mykkanen L, Tracy RP, Haffner SM. Chronic subclinical inflammation as part of the insulin resistance syndrome: the Insulin Resistance Atherosclerosis Study (IRAS). Circulation. 2000 Jul 4;102(1):42-7. doi: 10.1161/01.cir.102.1.42. PMID 10880413
- [Background] Dandona P, Chaudhuri A, Ghanim H, Mohanty P. Insulin as an anti-inflammatory and antiatherogenic modulator. J Am Coll Cardiol. 2009 Feb 3;53(5 Suppl):S14-20. doi: 10.1016/j.jacc.2008.10.038. PMID 19179212
- [Background] Dogne JM, Hanson J, Pratico D. Thromboxane, prostacyclin and isoprostanes: therapeutic targets in atherogenesis. Trends Pharmacol Sci. 2005 Dec;26(12):639-44. doi: 10.1016/j.tips.2005.10.001. Epub 2005 Oct 21. PMID 16243403
- [Background] Buscemi S, Verga S, Cottone S, Azzolina V, Buscemi B, Gioia D, Cerasola G. Glycaemic variability and inflammation in subjects with metabolic syndrome. Acta Diabetol. 2009 Mar;46(1):55-61. doi: 10.1007/s00592-008-0061-8. Epub 2008 Sep 26. PMID 18818862
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Ceriello A, Esposito K, Piconi L, Ihnat MA, Thorpe JE, Testa R, Boemi M, Giugliano D. Oscillating glucose is more deleterious to endothelial function and oxidative stress than mean glucose in normal and type 2 diabetic patients. Diabetes. 2008 May;57(5):1349-54. doi: 10.2337/db08-0063. Epub 2008 Feb 25. PMID 18299315
- [Background] Esposito K, Ciotola M, Carleo D, Schisano B, Sardelli L, Di Tommaso D, Misso L, Saccomanno F, Ceriello A, Giugliano D. Post-meal glucose peaks at home associate with carotid intima-media thickness in type 2 diabetes. J Clin Endocrinol Metab. 2008 Apr;93(4):1345-50. doi: 10.1210/jc.2007-2000. Epub 2008 Jan 15. PMID 18198229
- [Background] Esposito K, Giugliano D, Nappo F, Marfella R; Campanian Postprandial Hyperglycemia Study Group. Regression of carotid atherosclerosis by control of postprandial hyperglycemia in type 2 diabetes mellitus. Circulation. 2004 Jul 13;110(2):214-9. doi: 10.1161/01.CIR.0000134501.57864.66. Epub 2004 Jun 14. PMID 15197140
- [Background] Stehouwer CD, Gall MA, Twisk JW, Knudsen E, Emeis JJ, Parving HH. Increased urinary albumin excretion, endothelial dysfunction, and chronic low-grade inflammation in type 2 diabetes: progressive, interrelated, and independently associated with risk of death. Diabetes. 2002 Apr;51(4):1157-65. doi: 10.2337/diabetes.51.4.1157. PMID 11916939
- [Background] Shikano M, Sobajima H, Yoshikawa H, Toba T, Kushimoto H, Katsumata H, Tomita M, Kawashima S. Usefulness of a highly sensitive urinary and serum IL-6 assay in patients with diabetic nephropathy. Nephron. 2000 May;85(1):81-5. doi: 10.1159/000045634. PMID 10773760
- [Background] KDOQI. KDOQI Clinical Practice Guidelines and Clinical Practice Recommendations for Diabetes and Chronic Kidney Disease. Am J Kidney Dis. 2007 Feb;49(2 Suppl 2):S12-154. doi: 10.1053/j.ajkd.2006.12.005. No abstract available. PMID 17276798
- [Background] Dinneen SF, Gerstein HC. The association of microalbuminuria and mortality in non-insulin-dependent diabetes mellitus. A systematic overview of the literature. Arch Intern Med. 1997 Jul 14;157(13):1413-8. PMID 9224218
- [Background] Gerstein HC, Mann JF, Yi Q, Zinman B, Dinneen SF, Hoogwerf B, Halle JP, Young J, Rashkow A, Joyce C, Nawaz S, Yusuf S; HOPE Study Investigators. Albuminuria and risk of cardiovascular events, death, and heart failure in diabetic and nondiabetic individuals. JAMA. 2001 Jul 25;286(4):421-6. doi: 10.1001/jama.286.4.421. PMID 11466120
- [Background] Ruggenenti P, Remuzzi G. Time to abandon microalbuminuria? Kidney Int. 2006 Oct;70(7):1214-22. doi: 10.1038/sj.ki.5001729. Epub 2006 Jul 26. PMID 16871239
- [Background] Calle EE, Rodriguez C, Walker-Thurmond K, Thun MJ. Overweight, obesity, and mortality from cancer in a prospectively studied cohort of U.S. adults. N Engl J Med. 2003 Apr 24;348(17):1625-38. doi: 10.1056/NEJMoa021423. PMID 12711737
- [Background] Robinson RT, Harris ND, Ireland RH, Lee S, Newman C, Heller SR. Mechanisms of abnormal cardiac repolarization during insulin-induced hypoglycemia. Diabetes. 2003 Jun;52(6):1469-74. doi: 10.2337/diabetes.52.6.1469. PMID 12765959
- [Background] Desouza C, Salazar H, Cheong B, Murgo J, Fonseca V. Association of hypoglycemia and cardiac ischemia: a study based on continuous monitoring. Diabetes Care. 2003 May;26(5):1485-9. doi: 10.2337/diacare.26.5.1485. PMID 12716809
- [Background] Gill GV, Woodward A, Casson IF, Weston PJ. Cardiac arrhythmia and nocturnal hypoglycaemia in type 1 diabetes--the 'dead in bed' syndrome revisited. Diabetologia. 2009 Jan;52(1):42-5. doi: 10.1007/s00125-008-1177-7. Epub 2008 Oct 30. PMID 18972096
- [Background] Dungan KM, Buse JB, Largay J, Kelly MM, Button EA, Kato S, Wittlin S. 1,5-anhydroglucitol and postprandial hyperglycemia as measured by continuous glucose monitoring system in moderately controlled patients with diabetes. Diabetes Care. 2006 Jun;29(6):1214-9. doi: 10.2337/dc06-1910. PMID 16731998
- [Background] Kadowaki T, Yamauchi T. Adiponectin and adiponectin receptors. Endocr Rev. 2005 May;26(3):439-51. doi: 10.1210/er.2005-0005. PMID 15897298
- [Background] Sun J, Xu Y, Deng H, Sun S, Dai Z, Sun Y. Intermittent high glucose exacerbates the aberrant production of adiponectin and resistin through mitochondrial superoxide overproduction in adipocytes. J Mol Endocrinol. 2010 Mar;44(3):179-85. doi: 10.1677/JME-09-0088. PMID 20154025
- [Background] Bergt C, Pennathur S, Fu X, Byun J, O'Brien K, McDonald TO, Singh P, Anantharamaiah GM, Chait A, Brunzell J, Geary RL, Oram JF, Heinecke JW. The myeloperoxidase product hypochlorous acid oxidizes HDL in the human artery wall and impairs ABCA1-dependent cholesterol transport. Proc Natl Acad Sci U S A. 2004 Aug 31;101(35):13032-7. doi: 10.1073/pnas.0405292101. Epub 2004 Aug 23. PMID 15326314
- [Background] Shao B, Pennathur S, Pagani I, Oda MN, Witztum JL, Oram JF, Heinecke JW. Modifying apolipoprotein A-I by malondialdehyde, but not by an array of other reactive carbonyls, blocks cholesterol efflux by the ABCA1 pathway. J Biol Chem. 2010 Jun 11;285(24):18473-84. doi: 10.1074/jbc.M110.118182. Epub 2010 Apr 8. PMID 20378541
- [Background] Vaisar T, Pennathur S, Green PS, Gharib SA, Hoofnagle AN, Cheung MC, Byun J, Vuletic S, Kassim S, Singh P, Chea H, Knopp RH, Brunzell J, Geary R, Chait A, Zhao XQ, Elkon K, Marcovina S, Ridker P, Oram JF, Heinecke JW. Shotgun proteomics implicates protease inhibition and complement activation in the antiinflammatory properties of HDL. J Clin Invest. 2007 Mar;117(3):746-56. doi: 10.1172/JCI26206. PMID 17332893
- [Background] Green PS, Vaisar T, Pennathur S, Kulstad JJ, Moore AB, Marcovina S, Brunzell J, Knopp RH, Zhao XQ, Heinecke JW. Combined statin and niacin therapy remodels the high-density lipoprotein proteome. Circulation. 2008 Sep 16;118(12):1259-67. doi: 10.1161/CIRCULATIONAHA.108.770669. Epub 2008 Sep 2. PMID 18765395
- [Background] Hoofnagle AN, Wu M, Gosmanova AK, Becker JO, Wijsman EM, Brunzell JD, Kahn SE, Knopp RH, Lyons TJ, Heinecke JW. Low clusterin levels in high-density lipoprotein associate with insulin resistance, obesity, and dyslipoproteinemia. Arterioscler Thromb Vasc Biol. 2010 Dec;30(12):2528-34. doi: 10.1161/ATVBAHA.110.212894. Epub 2010 Sep 16. PMID 20847305
- [Background] Rosenfeld SI, Packman CH, Leddy JP. Inhibition of the lytic action of cell-bound terminal complement components by human high density lipoproteins and apoproteins. J Clin Invest. 1983 Apr;71(4):795-808. doi: 10.1172/jci110833. PMID 6403580
- [Background] Imhof A, Charnay Y, Vallet PG, Aronow B, Kovari E, French LE, Bouras C, Giannakopoulos P. Sustained astrocytic clusterin expression improves remodeling after brain ischemia. Neurobiol Dis. 2006 May;22(2):274-83. doi: 10.1016/j.nbd.2005.11.009. Epub 2006 Feb 10. PMID 16473512
- [Background] Rosenberg ME, Girton R, Finkel D, Chmielewski D, Barrie A 3rd, Witte DP, Zhu G, Bissler JJ, Harmony JA, Aronow BJ. Apolipoprotein J/clusterin prevents a progressive glomerulopathy of aging. Mol Cell Biol. 2002 Mar;22(6):1893-902. doi: 10.1128/MCB.22.6.1893-1902.2002. PMID 11865066
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Tamborlane WV, Beck RW, Bode BW, Buckingham B, Chase HP, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Hirsch IB, Huang ES, Kollman C, Kowalski AJ, Laffel L, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer S, Wilson DM, Wolpert H, Wysocki T, Xing D. Continuous glucose monitoring and intensive treatment of type 1 diabetes. N Engl J Med. 2008 Oct 2;359(14):1464-76. doi: 10.1056/NEJMoa0805017. Epub 2008 Sep 8. PMID 18779236
- [Background] Service FJ, Molnar GD, Rosevear JW, Ackerman E, Gatewood LC, Taylor WF. Mean amplitude of glycemic excursions, a measure of diabetic instability. Diabetes. 1970 Sep;19(9):644-55. doi: 10.2337/diab.19.9.644. No abstract available. PMID 5469118
- [Background] Clarke W, Kovatchev B. Statistical tools to analyze continuous glucose monitor data. Diabetes Technol Ther. 2009 Jun;11 Suppl 1(Suppl 1):S45-54. doi: 10.1089/dia.2008.0138. PMID 19469677
- [Background] Kovatchev BP, Clarke WL, Breton M, Brayman K, McCall A. Quantifying temporal glucose variability in diabetes via continuous glucose monitoring: mathematical methods and clinical application. Diabetes Technol Ther. 2005 Dec;7(6):849-62. doi: 10.1089/dia.2005.7.849. PMID 16386091
- [Background] McDonnell CM, Donath SM, Vidmar SI, Werther GA, Cameron FJ. A novel approach to continuous glucose analysis utilizing glycemic variation. Diabetes Technol Ther. 2005 Apr;7(2):253-63. doi: 10.1089/dia.2005.7.253. PMID 15857227
- [Background] Hirsch IB. Blood glucose monitoring technology: translating data into practice. Endocr Pract. 2004 Jan-Feb;10(1):67-76. doi: 10.4158/EP.10.1.67. PMID 15251625
- [Background] Rodbard D. New and improved methods to characterize glycemic variability using continuous glucose monitoring. Diabetes Technol Ther. 2009 Sep;11(9):551-65. doi: 10.1089/dia.2009.0015. PMID 19764834
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Beck RW, Hirsch IB, Laffel L, Tamborlane WV, Bode BW, Buckingham B, Chase P, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Huang ES, Kollman C, Kowalski AJ, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer SA, Wilson DM, Wolpert H, Wysocki T, Xing D. The effect of continuous glucose monitoring in well-controlled type 1 diabetes. Diabetes Care. 2009 Aug;32(8):1378-83. doi: 10.2337/dc09-0108. Epub 2009 May 8. PMID 19429875
- [Background] Hirsch IB, Brownlee M. Beyond hemoglobin A1c--need for additional markers of risk for diabetic microvascular complications. JAMA. 2010 Jun 9;303(22):2291-2. doi: 10.1001/jama.2010.785. No abstract available. PMID 20530784
- [Background] Basevi V, Di Mario S, Morciano C, Nonino F, Magrini N. Comment on: American Diabetes Association. Standards of medical care in diabetes--2011. Diabetes Care 2011;34(Suppl. 1):S11-S61. Diabetes Care. 2011 May;34(5):e53; author reply e54. doi: 10.2337/dc11-0174. No abstract available. PMID 21525493
- [Result] FLAT-SUGAR Trial Investigators. Glucose Variability in a 26-Week Randomized Comparison of Mealtime Treatment With Rapid-Acting Insulin Versus GLP-1 Agonist in Participants With Type 2 Diabetes at High Cardiovascular Risk. Diabetes Care. 2016 Jun;39(6):973-81. doi: 10.2337/dc15-2782. Epub 2016 Apr 19. PMID 27208320
- [Derived] FLAT-SUGAR Trial Investigators; Probstfield JL, Hirsch I, O'Brien K, Davis B, Bergenstal R, Kingry C, Khakpour D, Pressel S, Branch KR, Riddle M. Design of FLAT-SUGAR: Randomized Trial of Prandial Insulin Versus Prandial GLP-1 Receptor Agonist Together With Basal Insulin and Metformin for High-Risk Type 2 Diabetes. Diabetes Care. 2015 Aug;38(8):1558-66. doi: 10.2337/dc14-2689. Epub 2015 Jun 11. PMID 26068865

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Glargine, Metformin, Exenatide: Drug: Insulin Glargine Glargine-injectable, variable, QD, 6 months Drug: Metformin Metformin-oral, up to 1000mg, BID, 6 months Drug: Exenatide Injectable, 5mcg, BID, 6 months
- Insulin Glargine, Metformin, Prandial Insulin: Drug: Insulin Glargine Glargine-injectable, variable, QD, 6 months Drug: Metformin Metformin-oral, up to 1000mg, BID, 6 months Drug: Prandial insulin Aspart or glulisine or lispro
Period: Overall Study
Arm/Group | Insulin Glargine, Metformin, Exenatide | Insulin Glargine, Metformin, Prandial Insulin
Started | 52 | 50
Completed | 49 | 47
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Pancreatic Cancer | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Insulin Glargine, Metformin, Exenatide: Approximately 60 Type 2 DM participants will be instructed on an AHA/ADA meal plan. Insulin Glargine, metformin and exenatide will used as a combination strategy to control individual HBA1Cs between 6.7 and 7.3% throughout the trial.
  "GLIPULIN:" [insulin glargine, metformin, exenatide (GLP-1-agonist)]: Glargine-injectable, variable, QD, 6 months Metformin-oral, up to 1000mg, BID, 6 months Exenatide-injectable, 5mcg, BID, 6 months
- Glargine, Metformin, Prandial Insulin: Approximately 60 type 2 DM participants will be instructed in AHA/ADA meal plan. Insulin Glargine, metformin and one of 3 prandial insulins will be used as combination strategy to control individual HBA1Cs between 6.7 and 7.3%. Prandial Insulins (aspart, glulisine or lispro)
  Insulin glargine, metformin, prandial insulin: Approximately 60 type 2 DM participants will be instructed in AHA/ADA meal plan. Insulin Glargine, metformin and one of 3 prandial insulins will be used as combination strategy to control individual HBA1Cs between 6.7 and 7.3%. Prandial Insulins (aspart, glulisine or lispro)
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine, Metformin, Exenatide | Glargine, Metformin, Prandial Insulin | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Customized [Mean (Standard Deviation); unit: years] | 62 (8) | 63 (7) | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 36 | 28 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 43 | 40 | 83
  Black, Non-Hispanic | 6 | 7 | 13
  Hispanic | 1 | 3 | 4
  Other | 2 | 0 | 2
Glycosylated hemoglobin (HbA1C) [Mean (Standard Deviation); unit: %] | 7.9 (0.3) | 7.9 (0.3) | 7.9 (0.4)
Median Duration of Diabetes [Median (Standard Deviation); unit: years] | 15 (9) | 16 (7) | 15 (8)
Previous Cardiovascular (CV) Event [Count of Participants; unit: Participants] | 20 | 14 | 34
Previous Congestive Heart Failure (CHF) [Count of Participants; unit: Participants] | 3 | 0 | 3
Weight [Mean (Standard Deviation); unit: kg] | 101.3 (14.2) | 99.7 (17.8) | 100.5 (16)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.2 (5.0) | 33.7 (5.1) | 33.9 (5.1)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 113.9 (16.6) | 112.8 (14.1) | 113.4 (15.4)
Blood Pressure- [Mean (Standard Deviation); unit: mmHg]
  Systolic | 131.7 (13.6) | 129.1 (15.2) | 130.4 (14.4)
  Diastolic | 73.5 (11.3) | 73.1 (9.8) | 73.3 (10.5)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 70.5 (10.5) | 72.4 (10.4) | 71.4 (10.4)
C-peptide [Mean (Standard Deviation); unit: nmol/L] | 0.80 (0.07) | 0.73 (0.10) | 0.77 (0.77)
Creatinine [Mean (Standard Deviation); unit: micro mol/L] | 79.56 (17.68) | 79.56 (17.68) | 79.56 (17.68)
Alanine Transaminase (ALT) [Mean (Standard Deviation); unit: micro kat/L] | 37.6 (22.8) | 32.4 (14.8) | 35.0 (19.3)
Albumin/Creatinine Ratio [Mean (Standard Deviation); unit: mg/gm] | 3.95 (7.83) | 4.92 (16.94) | 4.23 (13.05)
Glucose Lowering Medications (prescreening) [Count of Participants; unit: Participants]
  Insulin | 52 | 50 | 102
  Basal insulin only | 14 | 12 | 26
  Prandial Insulin only | 1 | 3 | 4
  Basal + 1 or more Prandial insulin | 32 | 29 | 61
  Premixed insulin 1 or 2 injections | 2 | 3 | 5
  Metformin | 46 | 45 | 91
  Secretagogue | 11 | 13 | 24
  Thiazolidinedione | 3 | 1 | 4
  Glucagon-like peptide-1 receptor agonist(GLP- 1RA) | 0 | 4 | 4
  Dipeptidyl peptidase-4 (DPP-4) inhibitor | 1 | 2 | 3
Glucose coefficient of variation (CV) [Mean (Standard Deviation); unit: percentage] — Coefficient of variation (CV) = Standard deviation glucose/Mean glucose x 100
  percentage | 31.9 (6.1) | 30.0 (6.1) | 31.0 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Variation at 26 Weeks Minus Coefficient of Variation at Baseline
Description: The change in the coefficient of variation (CV) of continuous glucose readings, as assessed by Continuous Glucose Monitoring (CGM)
Time Frame: At baseline, 6 months of intervention
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Insulin Glargine, Metformin, Exenatide: 52 randomized, 49 completed, 47 had complete data collection for primary endpoint
- Insulin Glargine, Metformin, Prandial Insulin: 50 randomized, 47 completed protocol, 45 had complete data analyzed for primary endpoint.
Arm/Group | Insulin Glargine, Metformin, Exenatide | Insulin Glargine, Metformin, Prandial Insulin
Number analyzed (Participants) | 47 | 45
percentage | -2.43 (7.89) | 0.44 (5.50)
Statistical Analysis 1: Comparison: Insulin Glargine, Metformin, Exenatide vs Insulin Glargine, Metformin, Prandial Insulin; Two-tailed t test with type I error = 0.05, a sample of 110 participants (55 per group) would give 90% power to detect a difference of a mean change from baseline of 5 CV units (SD = 8) between control and treatment groups. An ANCOVA model, adjusting for baseline value and clinical site, was to be performed. If residual values from the ANCOVA indicated nonnormality in distribution by Shapiro-Wilk testing, a Wilcoxon rank sum test was used instead; Test type: Superiority; p < 0.024, Wilcoxon (Mann-Whitney) — Wilcoxon rank sum test was used due to nonnormality distribution; Wilcoxon

2. Secondary Outcome: Number of Participants With Hypoglycemia
Description: Severe hypoglycemia-documented glucose <50mg/dl (participant journal), and hypoglycemic attacks requiring hospitalization, or treatment by emergency personnel.
Time Frame: 26 weeks
Population: All participants that completed were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Insulin Glargine, Metformin, Exenatide: 52 randomized, 49 completed,
- Insulin Glargine, Metformin, Prandial Insulin: 50 randomized, 47 completed protocol,
Arm/Group | Insulin Glargine, Metformin, Exenatide | Insulin Glargine, Metformin, Prandial Insulin
Number analyzed (Participants) | 49 | 47
Participants | 0 | 0

3. Secondary Outcome: Weight Change During Trial
Description: Weight in kg at 26 weeks minus weight at baseline.
Time Frame: Baseline vs 26 weeks
Population: Participants with valid weights at baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Insulin Glargine, Metformin, Exenatide: 52 randomized, 49 completed
- Insulin Glargine, Metformin, Prandial Insulin: 50 randomized, 47 completed protocol
Arm/Group | Insulin Glargine, Metformin, Exenatide | Insulin Glargine, Metformin, Prandial Insulin
Number analyzed (Participants) | 45 | 45
kg | -4.8 (3.3) | 0.7 (3.3)
Statistical Analysis 1: Comparison: Insulin Glargine, Metformin, Exenatide vs Insulin Glargine, Metformin, Prandial Insulin; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

4. Other Pre Specified Outcome: HbA1C Levels
Description: % of glycosylated hemoglobin in whole blood at 26 weeks
Time Frame: Baseline vs 26 weeks
Measure: Mean (Standard Deviation); unit: % of HbA1C
Groups:
- Insulin Glargine, Metformin, Exenatide: 52 randomized, 49 completed, 45 had complete data collection for secondary endpoint
- Insulin Glargine, Metformin, Prandial Insulin: 50 randomized, 47 completed protocol, 45 had complete data analyzed for secondary endpoint.
Arm/Group | Insulin Glargine, Metformin, Exenatide | Insulin Glargine, Metformin, Prandial Insulin
Number analyzed (Participants) | 45 | 45
% of HbA1C | 7.1 (0.6) | 7.2 (0.6)
Statistical Analysis 1: Comparison: Insulin Glargine, Metformin, Exenatide vs Insulin Glargine, Metformin, Prandial Insulin; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 34- 36 weeks
Arm/Group | Insulin Glargine, Metformin, Exenatide | Insulin Glargine, Metformin, Prandial Insulin
All-Cause Mortality (participants affected / at risk) | 1/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 4/52 | 5/50
Other Adverse Events (participants affected / at risk) | 46/52 | 37/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine, Metformin, Exenatide (N=52) | Insulin Glargine, Metformin, Prandial Insulin (N=50)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Stapedotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Human anaplasmosis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine, Metformin, Exenatide (N=52) | Insulin Glargine, Metformin, Prandial Insulin (N=50)
Sinus arrest (Cardiac disorders) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 2 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (3) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 3 (4) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 20 (20) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Local reaction (General disorders) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 2 (3)
Infusion site bruising (General disorders) | 0 (0) | 1 (1)
Application site burn (General disorders) | 1 (1) | 0 (0)
Device capturing issue (General disorders) | 2 (2) | 1 (1)
Circumstance or information capable of leading to device use error (General disorders) | 0 (0) | 1 (1)
Administration site erythema (General disorders) | 1 (1) | 0 (0)
Abcess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cojunctiviris (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 5 (5)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compensatory sweating (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menopausal disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 5 (7) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Metatarsal excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Antiinflammatory therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes